CLINICAL TRIAL: NCT02497027
Title: Pharmacogenetic Testing in an Outpatient Population of Patients With Major Depressive Disorder or Depressive Disorder Not Otherwise Specified
Brief Title: Pharmacogenetic Testing in an Outpatient Population of Patients With Depression
Acronym: PGx-UPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AIHG-1440-PGxUPA
Record Dates: First submitted 2015-06-15; First posted 2015-07-14 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Depression
Keywords: pharmacogenetic, pharmacogenomic, depressive, mental health
MeSH Terms: conditions — Depression; Psychological Well-Being | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 4-Week Group (Other): Pharmacogenetic testing released to physician at 4 weeks following enrollment into study
  Interventions: Other: pharmacogenetic testing
- 12-Week Group (Other): Pharmacogenetic testing released to physician at 12 weeks following enrollment into study
  Interventions: Other: pharmacogenetic testing

INTERVENTIONS:
Other: pharmacogenetic testing — pharmacogenetic testing report released to physician at 4 weeks post enrollment
  Arms: 4-Week Group
Other: pharmacogenetic testing — pharmacogenetic testing report released to physician at 12 weeks post enrollment
  Arms: 12-Week Group

SUMMARY:
This is a randomized, control group design of pharmacogenetic implementation in a mental health population of subjects taking anti-depressants and/or anti-psychotics with a new or current primary or secondary diagnosis of Major Depressive Disorder (MDD) or Depressive Disorder Not Otherwise Specified (DDNOS).

DETAILED DESCRIPTION:
This is a randomized, control group design of pharmacogenetic implementation in a mental health population of subjects taking anti-depressants and/or anti-psychotics with a new or current primary or secondary diagnosis of Major Depressive Disorder (MDD) or Depressive Disorder Not Otherwise Specified (DDNOS). Prospective data will be collected on all subjects until study completion at 24-25 weeks post enrollment. Claims data may be reviewed per pay, if such data are readily available in a timely manner.

ELIGIBILITY:
Inclusion Criteria:

* Current primary or secondary diagnosis of Major Depressive Disorder or Depressive Disorder Not Otherwise Specified
* Have moderate to severe depression as identified by PHQ-9 scoring of 10 or greater
* Taking or be newly prescribed an anti-depressant or anti-psychotic medication
* Able to provide informed consent
* Prescribing physician practices at the Avera Medical Group University Psychiatry Associates clinic in Sioux Falls, SD

Exclusion Criteria:

* Pregnant or breastfeeding
* Active and/or unstable diagnosis of substance abuse, excluding nicotine
* Primary diagnosis of dementia, bipolar disorder (any type), schizophrenia, schizoaffective disorder, or personality disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-02; Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Depression score | 24 weeks
  response to medication following medication recommendation guided by pharmacogenetic testing

SECONDARY OUTCOMES:
Clinical utility questionnaire | 24 weeks
  This will be assessed through review of medical records and a study compliance questionnaire to be completed by the prescribing physician

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Stanley, MD, Principal Investigator — Avera McKennan Hospital & University Health Center
Locations (1):
- Avera McKennan Hospital & University Health Center, Sioux Falls, South Dakota, United States